CLINICAL TRIAL: NCT00056394
Title: Coping Skills Training for Early Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: Pro00007830; R01AR047218 (NIH); NIAMS-086
Record Dates: First submitted 2003-03-11; First posted 2003-03-12 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2013-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Early Rheumatoid Arthritis; Coping Skills Training; Pain; Physical Disability; Psychological Disability; Daily Diary Measures
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive comprehensive pain coping skills.
  Interventions: Behavioral: Comprehensive Coping Skills Training
- 2 (Active Comparator): Participants will receive arthritis education.
  Interventions: Behavioral: Arthritis Education Sessions
- 3 (Active Comparator): Participants will receive standard care.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Comprehensive Coping Skills Training — 10 weekly, 80-minute coping skills treatment sessions, followed by a series of six biweekly follow-up telephone calls.
  Arms: 1
Behavioral: Arthritis Education Sessions — 10 weekly, 80-minute treatment sessions, followed by a series of six biweekly follow-up telephone calls. Participants will learn about the nature and treatment of rheumatoid arthritis as well as the benefits of exercise and joint protection.
  Arms: 2
Behavioral: Standard Care — Usual care from participants' rheumatologists but no treatment sessions.
  Arms: 3

SUMMARY:
Rheumatoid arthritis (RA) is the most common inflammatory arthritis and a major health problem. Medical treatments are now being used much earlier in the course of RA, but these treatments do not address the challenges of coping with the early stages of this disease. This study will determine whether a comprehensive coping skills training program can decrease pain, psychological disability, and physical disability in patients with early RA.

DETAILED DESCRIPTION:
RA is a serious and complex disease that taxes patients' coping resources. Patients with RA must cope with pain and with major life stresses, including disruptions in their health, work, family, and marital functioning.

Recognition of the morbidity and mortality associated with RA has increased interest in early interventions. Rapid disease progression during the first few years of RA taxes patients' coping efforts. Those who cope well with the early stages of RA can maintain an active and rewarding lifestyle. Those who do not may become depressed, decrease physical activity, and develop a sedentary, restricted lifestyle that contributes to long-term disability and overdependence on family and friends.

This study will evaluate the effectiveness of early coping skills training (CST) to enhance self-efficacy, prepare patients to cope with future pain, and prevent the development of behaviors that may increase long-term psychological distress and physical disability. The comprehensive CST intervention combines traditional CST with CST components tailored to rheumatoid arthritis patients. It is designed to teach traditional coping skills such as attention diversion, cognitive restructuring, and changes in activity to control and decrease pain.

Participants will be randomized to one of three study groups: 1) comprehensive pain coping skills training; 2) arthritis education; or 3) standard care. Study participants assigned to the comprehensive CST and the arthritis education groups will be asked to attend ten weekly, 80-minute treatment sessions. These ten sessions will be followed by a series of six biweekly follow-up telephone calls.

Study participants in the arthritis education group will learn about the nature and treatment of rheumatoid arthritis as well as the benefits of exercise and joint protection. Study participants in the standard care group will continue to receive care from their rheumatologists but will not participate in any treatment sessions.

Measures of pain, disability, pain coping, and self efficacy will be collected during evaluation sessions before and after the treatment phase. Participants attend 5 evaluation sessions and will be followed for 18 months.

ELIGIBILITY:
Inclusion Criteria

* Meet at least 4 of the 7 criteria for RA classification based on the 1987 American College of Rheumatology criteria
* Onset of RA symptoms within 2 years of study entry

Exclusion Criteria

* Known organic disease that significantly affects function
* Rheumatic disorders in addition to RA that significantly affect function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2003-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Pain | Measured at Week 10
Psychological disability | Measured at Week 10
Physical disability | Measured at Week 10

SECONDARY OUTCOMES:
Erythrocyte sedimentation rate | Measured at Week 10
Joint tenderness count | Measured at Week 10
Grip strength | Measured at Week 10
Physician assessment of disease activity | Measured at Week 10
C reactive protein | Measured at Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Francis J. Keefe, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina